CLINICAL TRIAL: NCT02153827
Title: Shoulder External Rotator Eccentric Training for Subacromial Impingement Syndrome
Brief Title: Shoulder Eccentric External Rotator Training for Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: University of St. Augustine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12111308exp
Record Dates: First submitted 2014-03-31; First posted 2014-06-03 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2015-04

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder; Eccentric Training; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric External rotator training (Experimental): Eccentric Shoulder External Rotators along with scapular retraction and posterior shoulder stretching exercises.
  Interventions: Other: Eccentric Shoulder External Rotator Training
- General shoulder exercise (Sham Comparator): General shoulder exercise protocol of active flexion, abduction, scapular retraction and posterior shoulder stretching exercises.
  Interventions: Other: General Shoulder exercise

INTERVENTIONS:
Other: Eccentric Shoulder External Rotator Training — Eccentric training exercise for the external rotators, 3 sets of 15 daily.
  Arms: Eccentric External rotator training
Other: General Shoulder exercise — general exercise consisting of active shoulder movements
  Arms: General shoulder exercise

SUMMARY:
The purpose of this study is to examine the effects of eccentric exercise to the shoulder muscles for people with shoulder pain. Identifying specific exercise protocols for individuals with shoulder pain will provide evidence to help clinicians select the best interventions.

DETAILED DESCRIPTION:
Prior investigations for eccentric training of the shoulder have primarily utilized a pain provocation model for exercise progression. This method of progressing resistance training load and volume assumes that pain must be increased during the exercise movement for clinical benefit to occur. When the individual reports a reduction in pain, load is increased so that the provoking pain level returns. The contrast to this approach would be a performance based progression as utilized in the Blume et al study for shoulder eccentric training. This method progresses a patient based on ability to perform a higher number of repetitions at a given load without increasing symptoms which could be favorable in many clinical settings.

Further investigation on the role of eccentric training, specifically to the shoulder external rotators, in patients with SAPS is warranted. Thus, the aim of this investigation was to compare outcomes, for individuals diagnosed with SAPS, performing a six week protocol of eccentric training to the shoulder external rotators compared to a general exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Presence of non-acute shoulder pain (greater than 3 months duration)
* 3 out of the 6 following tests positive, Neer impingement, Hawkins-Kennedy impingement, empty can test, resisted external rotation test, palpable tenderness at the insertion of the supraspinatus or infraspinatus, and painful arc from 60° to 120° during active abduction.
* Age over 18 years old
* Sufficient ability to read English as required for completing questionnaires

Exclusion Criteria:

* Red flags noted in the patient's Medical Screening Questionnaire (MSQ) (ie. tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, prolonged history of steroid use)
* Full thickness supraspinatus or infraspinatus tendon tear as determined by a positive drop arm test, lag sign or rent test.
* Shoulder adhesive capsulitis as evidenced by a limitation in passive motion for all shoulder planes of movement.
* Having an upper extremity amputation.
* Individuals having a history of surgery to the cervical spine or involved upper extremity for a musculoskeletal, neurological or dermatological condition for which they are at the time of data collection receiving post-operative care.
* Pending legal action regarding their shoulder pain
* Inability to comply with treatment and follow up schedule
* Insufficient English language skills to complete all questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morey Kolber, PhD, PT, Study Chair — Nova Southeastern
Locations (1):
- University of St. Augustine, Saint Augustine, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588
- [Result] Camargo PR, Avila MA, Alburquerque-Sendin F, Asso NA, Hashimoto LH, Salvini TF. Eccentric training for shoulder abductors improves pain, function and isokinetic performance in subjects with shoulder impingement syndrome: a case series. Rev Bras Fisioter. 2012 Jan-Feb;16(1):74-83. doi: 10.1590/s1413-35552012000100013. PMID 22441232
- [Result] Maenhout AG, Mahieu NN, De Muynck M, De Wilde LF, Cools AM. Does adding heavy load eccentric training to rehabilitation of patients with unilateral subacromial impingement result in better outcome? A randomized, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1158-67. doi: 10.1007/s00167-012-2012-8. Epub 2012 May 12. PMID 22581193
- [Result] Bernhardsson S, Klintberg IH, Wendt GK. Evaluation of an exercise concept focusing on eccentric strength training of the rotator cuff for patients with subacromial impingement syndrome. Clin Rehabil. 2011 Jan;25(1):69-78. doi: 10.1177/0269215510376005. Epub 2010 Aug 16. PMID 20713438
- [Result] Jonsson P, Wahlstrom P, Ohberg L, Alfredson H. Eccentric training in chronic painful impingement syndrome of the shoulder: results of a pilot study. Knee Surg Sports Traumatol Arthrosc. 2006 Jan;14(1):76-81. doi: 10.1007/s00167-004-0611-8. Epub 2005 May 5. PMID 15877219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2014 - October 2015 participants were recruited from the local community via publicly displayed flyers.
Pre-assignment Details: none to report
Groups:
- Eccentric External Rotator Training: Eccentric Shoulder External Rotator Training
Period: Overall Study
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Started | 25 | 23
Completed | 22 | 14
Not Completed | 3 | 9
Not completed — Lost to Follow-up | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.35 (17.88) | 48.35 (16.89) | 45.85 (17.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 15 | 13 | 28
Body mass [Mean (Standard Deviation); unit: Kilograms] | 79.87 (15.04) | 81.90 (18.55) | 80.88 (16.795)

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario Rotator Cuff Index
Description: shoulder functional self report measure is a disease specific self reported outcome measure for individuals experiencing rotator cuff pathology. A score of 0 is the minimum score and indicates low levels of shoulder function. A score of 100 is the maximum score and indicates full shoulder function. Scores are derived by summing all 5 subscales and dividing that number by the total available number of 2100. Units for each item are derived from a visual analog scale totaling 100cm.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale derived from 100cm vas
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Number analyzed (Participants) | 22 | 14
units on a scale derived from 100cm vas | 92.72 (8.98) | 77.15 (15.91)

2. Secondary Outcome: Global Rating of Change
Description: Global rating of change is a single item questionnaire asking about total change since beginning treatment. The scale ranges from -7 (a great deal worse) to +7 (a great deal better). The unit of measure is scores on a scale.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Number analyzed (Participants) | 22 | 14
units on a scale | 5.00 (2.25) | 2.50 (2.65)

3. Secondary Outcome: Numeric Pain Rating Scale
Description: 0-10 pain scale with 0 meaning no pain and 10 being maximal pain. This is derived from a single item questionnaire.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Number analyzed (Participants) | 22 | 14
units on a scale 0-10 | 1.04 (1.62) | 2.14 (1.83)

4. Secondary Outcome: Shoulder Active Range of Motion
Description: Degrees of shoulder elevation with 0 being the least and 180 being the greatest.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Number analyzed (Participants) | 22 | 14
Degrees | 175 (11) | 170 (15)

5. Secondary Outcome: Upper Quarter Y Balance Test
Description: Measure of single arm reach with 0 being the least and higher numbers indicating greater distance reached.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm of reach divided by limb length
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Number analyzed (Participants) | 22 | 14
cm of reach divided by limb length | 1.21 (13) | 1.12 (.29)

ADVERSE EVENTS:
Time Frame: the 6 months during study data collection for each participant
Arm/Group | Eccentric External Rotator Training | General Shoulder Exercise
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No